CLINICAL TRIAL: NCT02736760
Title: Prospective, Randomized, Controlled, Multicenter, Two-armed, Study Comparing Daylight Photodynamic Therapy Using MAL With Cryosurgery for the Treatment and Prophylaxis of Actinic Keratoses in Photodamaged Skin of the Face
Brief Title: Daylight-PDT With MAL for AK and Photodamaged Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Professor Dr. Sigrid Karrer, Professor, University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daylight_01
Record Dates: First submitted 2016-03-11; First posted 2016-04-13 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Actinic Keratoses; Photodamaged Skin
MeSH Terms: conditions — Keratosis, Actinic | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daylight photodynamic therapy (PDT) (Experimental): One intervention in the daylight photodynamic therapy arm:
  Daylight photodynamic therapy using Methylaminolevulinate (MAL) will be performed five times within 18 months (visits 1-5). In the PDT group the patients will apply a chemical sunscreen (SPF 50+) to the whole face and other light-exposed, unprotected areas of the skin. After at least 15 minutes a lesion preparation of AKs (removal of crusts) will be performed and methylaminolevulinate (MAL) will be applied in a thin layer to the whole face. Within 30 min after MAL application patients expose themselves to daylight for 2 hours.
  Interventions: Drug: Daylight photodynamic therapy using Methylaminolevulinate (MAL)
- Cryosurgery (Active Comparator): In the control group, cryosurgery will be performed at visit 1, and in case of non-cleared or newly occurred AKs at visits 2-5. In the control group, cryosurgery will be performed using liquid nitrogen spray in each AK lesion; this will be done at visit 1 and, if necessary, also at visits 2-5. At visits 2-6, the efficacy of the treatment will be evaluated by the observer by documenting all existing and newly appearing AKs in the face.
  Interventions: Procedure: Cryosurgery

INTERVENTIONS:
Drug: Daylight photodynamic therapy using Methylaminolevulinate (MAL) — In the Daylight photodynamic therapy arm the patients will apply a sunscreen to the whole face which is followed by lesion preparation of AKs. Following this, MAL will be applied in a thin layer to the whole face. Within 30 min after MAL application patients expose themselves to daylight for 2 hours.
  5 photodynamic therapy treatment sessions (visits 1-5) will be performed within 18 months.
  Other Names: Daylight-PDT
  Arms: Daylight photodynamic therapy (PDT)
Procedure: Cryosurgery — In the control group, cryosurgery as standard reference therapy will be performed at visit 1, and in case of non-cleared or newly occurred AKs at visits 2-5. Cryosurgery of AK lesions will be investigated as standard reference therapy. Single freeze-thaw cryosurgery is performed using an open spraying procedure with liquid nitrogen with nozzle size C. After formation of an ice-ball of the required size, freeze time starts. Freeze time should lie between 5 s and 10 s.
  Arms: Cryosurgery

SUMMARY:
This study is a multicenter study investigating the clinical efficacy of repetitive daylight-PDT with MAL (Methylaminolevulinate) compared to cryosurgery in regard to prophylaxis and treatment of AKs (actinic keratoses) in the face. Patients will be randomly allocated to treatment groups. 5 PDT (photodynamic therapy) treatment sessions (visits 1-5) will be performed within 18 months. In the control group, cryosurgery will be performed at visit 1, and in case of non-cleared or newly occurred AKs at visits 2-5.

In the PDT group the patients will apply a chemical sunscreen (SPF 50+) to the whole face and other light-exposed, unprotected areas of the skin. After at least 15 minutes a lesion preparation of AKs (removal of crusts) will be performed and MAL will be applied in a thin layer to the whole face. Within 30 min after MAL application patients expose themselves to daylight for 2 hours. In the control group, cryosurgery will be performed using liquid nitrogen spray in each AK lesion; this will be done at visit 1 and, if necessary, also at visits 2-5. At visits 2-6, the efficacy of the treatment will be evaluated by the observer by documenting all existing and newly appearing AKs in the face.

DETAILED DESCRIPTION:
This study is a multicenter study investigating the clinical efficacy of repetitive daylight-PDT with MAL compared to cryosurgery in regard to prophylaxis and treatment of AKs in the face. Patients will be randomly allocated to treatment groups. 5 PDT treatment sessions (visits 1-5) will be performed within 18 months. In the control group, cryosurgery will be performed at visit 1, and in case of non-cleared or newly occurred AKs at visits 2-5.

Before application of the photosensitizer, an organic sunscreen (Actinica® lotion, LSF 50+) without mineral filters will be applied In the entire face.

After an absorption time of approximately 15 minutes and before applying MAL (Metvix®), the surface of the AK lesions will be prepared gently with a curette or a scalpel to remove scales and crusts and roughen the surface of the AK-lesions. This is to facilitate penetration of the cream and light to the AK lesions.

After lesion preparation, MAL (Metvix®) will be uniformly applied on the whole face in a thin layer.

Within 30 min after MAL application the patients go outside and expose themselves for 2 hours to daylight. Daylight-PDT can be performed from March until October, during non-rainy weather with an outdoor temperature of at least 10° Celsius. Daylight exposure must start at least 3 hours before sunset.

At the end of the exposure, residual photosensitizer is washed off and the patients spend the rest of the day indoors.

Cryosurgery of AK lesions will be investigated as standard reference therapy. Single freeze-thaw cryosurgery is performed using an open spraying procedure with liquid nitrogen with nozzle size C. After formation of an ice-ball of the required size, freeze time starts. Freeze time should lie between 5 s and 10 s.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been signed prior to or at Screening Visit
* Male and female patients with Fitzpatrick skin type I-IV
* Age > 40 years
* Negative pregnancy test in women of childbearing age
* Women in child-bearing age using highly efficient contraceptive methods (<1% failure rate per year)
* Clinical diagnosis of actinic keratosis (AK)
* A minimum of five non-hyperkeratotic, non-pigmented AK lesions in the face.
* Glogau Photodamage Classification Type II (moderate) - IV (severe)

Exclusion Criteria:

* Diagnosis of porphyria
* Hyperkeratotic or pigmented AK in the face
* Malignant skin tumors in the face or on the capillitium, requiring treatment
* Patients with clinically relevant suppression of the immune system (e.g. drug induced, infection) or organ transplant patients
* Pregnancy or lactation
* Planned aesthetic treatments in the face in the next 24 months (filler, peeling, botulinumtoxin, skin resurfacing)
* Known intolerance or allergy to MAL or to any other ingredient of Metvix® 160mg/g cream
* Known intolerance to Actinica® lotion
* Photosensitivity
* Suspected lack of compliance (e.g. due to dementia)
* Simultaneous participation in another clinical study or participation in another clinical study in the 30 days directly preceding inclusion
* Concomitant UV-phototherapy
* Skin diseases that might interfere with response evaluation of study treatment
* Skin sun sensitivity type V or VI according to Fitzpatrick
* PDT in the face during 6 months preceding study treatment
* Non-permitted medication:
* Topical treatment in the face during 4 weeks preceding study treatment with diclofenac, hydrochinone, peeling, 5-FU, ingenolmebutate, retinoids, podophyllin, azelaic acid, imiquimod or other agents, that could interfere with the evaluation of the efficacy of the study treatment, according to the investigator.
* Systemic treatment with retinoids
* Conditions that might interfere with the ability to understand the study and thus give written informed consent
* Rejuvenating treatments of the face during 3 months preceding study treatment, including filler, botulinumtoxin and IPL

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
The cumulative number of observed AKs at time points 2 to 6 (3 months after the first treatment to 24 months after the first treatment). | 24 months after the first treatment
  Newly occured AK lesions are counted at visit 2, visit 3, visit 4, visit 5 and visit 6.
  The number of newly occured AK lesions during the study are added up, therefore we included the term "cumulative".

SECONDARY OUTCOMES:
Complete clearance of AKs on lesion basis | This outcome measure is assessed three months after the first and the second treatment and 6 months after the third, fourth and fifth treatment.
  completely cleared AK lesions
  The first treatment ist performed at day 0 The second treatment is performed 3 months after the first treatment. The third treatment is performed 3 months after the second treatment. The fourth treatment is performed 6 months after the third treatment. The fifth treatment is performed 6 months after the fourth treatment.
Complete clearance of AKs on patient basis | This outcome measure is assessed three months after the first and the second treatment and 6 months after the third, fourth and fifth treatment.
  completely cleared AK lesions on patient basis
  The first treatment ist performed at day 0 The second treatment is performed 3 months after the first treatment. The third treatment is performed 3 months after the second treatment. The fourth treatment is performed 6 months after the third treatment. The fifth treatment is performed 6 months after the fourth treatment.
Photodamage parameters (fine lines, mottled pigmentation, tactile roughness, teleangiectasias, sallowness and global score for photoaging) will be evaluated on a 5-point scale according to Dover et al. | This outcome measure is assessed at day 0 (= the first treatment), three months after the first and the second treatment and 6 months after the third, fourth and fifth treatment.
  Photodamage parameters will be evaluated on a 5-point scale according to Dover et al. at all visits during the study
  The first treatment ist performed at day 0 (visit 1) The second treatment is performed 3 months after the first treatment (visit 2) The third treatment is performed 3 months after the second treatment (visit 3) The fourth treatment is performed 6 months after the third treatment (visit 4) The fifth treatment is performed 6 months after the fourth treatment (visit 5) The last visit is performed 6 months after the fifth treatment (visit 6)
Visual pain score | This outcome measure is assessed at day 0 (= the first treatment), three months after the first and the second treatment and 6 months after the third, fourth and fifth treatment
  For evaluation of tolerability of daylight-PDT and cryosurgery, a pain score (VAS) will be assessed and documented.
  The first treatment ist performed at day 0 (visit 1) The second treatment is performed 3 months after the first treatment (visit 2) The third treatment is performed 3 months after the second treatment (visit 3) The fourth treatment is performed 6 months after the third treatment (visit 4) The fifth treatment is performed 6 months after the fourth treatment (visit 5) The last visit is performed 6 months after the fifth treatment (visit 6)
Adverse events | This outcome measure is assessed at day 0 (= the first treatment), three months after the first and the second treatment and 6 months after the third, fourth and fifth treatment
  All adverse events and serious adverse events will be adequately documented.
  The first treatment ist performed at day 0 (visit 1) The second treatment is performed 3 months after the first treatment (visit 2) The third treatment is performed 3 months after the second treatment (visit 3) The fourth treatment is performed 6 months after the third treatment (visit 4) The fifth treatment is performed 6 months after the fourth treatment (visit 5) The last visit is performed 6 months after the fifth treatment (visit 6)
Patient satisfaction with cosmetic results | This outcome measure is assessed three months after day 0 and the second treatment and 6 months after the third, fourth and fifth treatment
  For evaluation of satisfaction with cosmetic results, patients and investigators fill in a standardized rating scale
  The first treatment ist performed at day 0 (visit 1) The second treatment is performed 3 months after the first treatment (visit 2) The third treatment is performed 3 months after the second treatment (visit 3) The fourth treatment is performed 6 months after the third treatment (visit 4) The fifth treatment is performed 6 months after the fourth treatment (visit 5) The last visit is performed 6 months after the fifth treatment (visit 6)
Skin-related quality of life | This outcome measure is assessed at day 0 and 24 months after day 0
  For evaluation of skin-related quality of life, study participants fill in the Dermatology Life Quality Index, a 10-item questionnaire for routine clinical use. Patients are asked about the impact of their AK and photodamaged skin and its treatment on their lives. Patients' quality of life is expressed in a single score ranging from 0 (no impact) to 30 (severe impact).

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - University hospital Regensburg, Regensburg, Bavaria
  - Hautzentrum Köln, Cologne
  - University Hospital Düsseldorf., Düsseldorf
  - Klinikum Vest GmbH Knappschaftskrankenhaus, Recklinghausen

REFERENCES:
- [Derived] Kohl E, Koller M, Zeman F, Szeimies RM, Philipp-Dormston WG, Prager W, Gerber PA, Karrer S. Daylight photodynamic therapy versus cryosurgery for the treatment and prophylaxis of actinic keratoses of the face - protocol of a multicenter, prospective, randomized, controlled, two-armed study. BMC Dermatol. 2017 Oct 25;17(1):12. doi: 10.1186/s12895-017-0064-7. PMID 29070025